CLINICAL TRIAL: NCT04731688
Title: A Weight Maintenance Program Promoting Fat Loss in Pregnancy in Women With Obesity
Acronym: Healthy Mamas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: California Polytechnic State University-San Luis Obispo (Other); Oregon Health and Science University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Leanne Redman, Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 2019-070; 1R01DK124806-01 (NIH)
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Gestational Weight Gain; Obesity
Keywords: Pregnancy; Body Composition
MeSH Terms: conditions — Gestational Weight Gain; Obesity

STUDY DESIGN:
Intervention Model Description: Two site randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be conducted by staff members who are masked to the participant's intervention group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight Maintenance Group (Experimental): Individuals in this group will receive all aspects of the Provider Directed Group plus a comprehensive behavioral fat mass loss intervention with food provision. Individuals in this group will be provided foods to eat to support weight maintenance and loss of body fat throughout pregnancy. They will be asked to attend two behavioral counseling sessions at the beginning of the study to help learn the program and set goals. They will return for brief visits with a lifestyle counselor every two weeks until 20 weeks gestation and at least once a month until delivery. Individuals will be provided a scale to help keep track of weight during pregnancy.
  Interventions: Behavioral: Weight Maintenance Group
- Provider Directed Group (No Intervention): Individuals in this group will receive what is standard practice by their prenatal care providers during pregnancy. In addition, individuals in this group will be asked to attend a brief session at the time of randomization to familiarize with the study and what is expected. They will also be provided with materials describing healthy behaviors in pregnancy.

INTERVENTIONS:
Behavioral: Weight Maintenance Group — The behavioral program is rooted in social learning theory and based on our existing prenatal intervention but with full food provision to ensure gestational fat mass loss is steady and closely supervised. Brief counseling sessions are designed to review self-monitoring records, reinforce adherence to the structured food provision program, problem-solve barriers, and provide additional support. Individuals will be provided with a structured meal plan designed to promote 25% calorie restriction during the second trimester followed by eucaloric intake during the 3rd trimester. Participants will be provided three meals and two snacks on 7 days at no cost.
  Arms: Weight Maintenance Group

SUMMARY:
The aims of this randomized controlled trial are to determine the effects of a lifestyle program that supports weight maintenance and fat mass loss during pregnancy in women with obesity on changes in 1) maternal weight, fat mass, and cardiometabolic risk factors; 2) safety measures, including fetal and neonatal growth; 3) the mediators and moderators of the fat mass loss intervention and 4) the effects gestational fat mass loss has on reducing incidence of adverse obstetrical outcomes, including non-elective cesarean delivery, gestational diabetes, hypertension, and pre-eclampsia.

DETAILED DESCRIPTION:
One hundred pregnant women with obesity who are otherwise healthy will be studied from early pregnancy until approximately 2 weeks postpartum. Major assessments will occur at baseline (13-16 weeks gestation), 27-29 weeks gestation, 35-37 weeks gestation, and approximately 2 weeks postpartum. Safety assessments will be collected every 4 weeks after enrollment. Participants will be randomized within site (approximately 50 individuals at Pennington Biomedical Research Center and approximately 50 individuals at California Polytechnic University) and obesity to either: Provider Directed Group or Weight Maintenance Group.

ELIGIBILITY:
Inclusion Criteria:

* Are pregnant less than or equal to 15 weeks gestation at screening
* Have a body mass index between 31.0 and 55.0 inclusive
* Have a confirmed viable singleton gestation
* Willing to receive randomization to either group
* Willing and able to eat the study foods
* Willing to enroll infant for study measurements after birth
* Receive clearance from the prenatal care provider for participation

Exclusion Criteria:

* Smoking, drug, or alcohol use
* Have a known fetal anomaly
* Have a non-pregnancy related illness
* Have pre-existing diabetes
* Have pre-existing hypertension
* Have severe anemia
* Have current mental health issue or eating disorder
* Short inter-pregnancy interval (<6 months since last pregnancy)
* Use of assisted reproductive technology
* Use of medications with known effects on body weight including over the counter medications and supplements for weight loss
* History of pre-eclampsia, prior small for gestational age infant, bariatric surgery
* Planning to move out of the area in the next 12 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 100 pregnant women with obesity will be enrolled.
Enrollment: 100 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Body weight | From study entry to approximately 2 weeks postpartum
  Body weight will be measured using a calibrated electrical scale with participants wearing a hospital gown and underwear.

SECONDARY OUTCOMES:
Fat mass | From study entry to approximately 2 weeks postpartum
  Fat mass will be assessed via a 3-compartment model in which fat mass is calculated from body weight, body density measured by the BODPOD, and total body water measured by deuterium dilution.

OTHER OUTCOMES:
Total body water | From study entry to approximately 2 weeks postpartum
  Total body water is assessed by deuterium dilution.
Fat-free mass | From study entry to approximately 2 weeks postpartum
  Fat-free mass will be calculated as the subtraction of fat mass from total body weight.
Fetal weight | From 19-22 weeks gestation to 39-42 weeks gestation
  Fetal weight is measured by ultrasound and estimated by Hadlock formula.
Infant body composition | Approximately 2 weeks old
  Infant body composition will be assessed via a 3-compartment model which includes body weight, PEAPOD, and dual-energy x-ray absorptiometry.
Dietary intake | From study entry to 35-37 weeks gestation
  Dietary intake is assessed by automated self-administered 24-hour dietary assessment tool (ASA-24).
Time Spent in Physical activity | From study entry to 35-37 weeks gestation
  Physical activity (amount of time spent in physical activity) is assessed by activPAL activity device over a period of 5-7 days.
Metabolic syndrome score | From study entry to approximately 2 weeks postpartum
  Metabolic syndrome score will be determined using measured blood pressure and waist circumference, and triglycerides, high density lipoprotein cholesterol, and glucose.
Perinatal outcomes | From study entry to approximately 2 weeks postpartum
  All perinatal outcomes (ie non-elective cesarean delivery, gestational diabetes, hypertension, pre-eclampsia) will be obtained by prenatal and delivery medical chart abstraction.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (2):
- United States (2):
  - California Polytechnic State University, San Luis Obispo, California
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Redman LM, Phelan S, Apolzan JW, Beyl RA, Altazan AD, Dickey MS, Simeon E, Flanagan EW, Cabre HE, Sparks JR, Kebbe M, Caughey AB, Valent AM, Hsia DS, Yin E, Keadle SK. Protocol for a randomised controlled trial of a weight maintenance intervention to promote fat loss in pregnant individuals with obesity. BMJ Open. 2025 Feb 25;15(2):e095804. doi: 10.1136/bmjopen-2024-095804. PMID 40000086